CLINICAL TRIAL: NCT05238025
Title: A Randomized, Double-blind, Phase 3 Trial to Assess Clinical Efficacy, Safety and Reactogenicity of the Recombinant MVA-BN® -RSV Vaccine in Adults ≥60 Years of Age
Brief Title: MVA-BN-RSV Vaccine Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated after the first RSV season because of the failure to meet the primary outcome measures of vaccine efficacy
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RSV-MVA-004
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Single dose MVA-BN-RSV (Experimental): Single dose (Week 0): MVA-BN-RSV virus with a titer of at least 3x10E8 Inf.U/0.5mL (intramuscular vaccination)
  Interventions: Biological: MVA-BN-RSV vaccine
- Group 2: Single dose Placebo (Experimental): Single dose of TBS (intramuscular injection; 0.5mL)
  Interventions: Biological: Tris Buffered Saline (TBS)

INTERVENTIONS:
Biological: MVA-BN-RSV vaccine — One injection, suspension for injection, intramuscular use, 0.5mL MVA-BN-RSV virus with a titer of at least 3 x 10E8 infectious units (Inf.U)/0.5mL in a Tris buffer at pH 7.7.
  Arms: Group 1: Single dose MVA-BN-RSV
Biological: Tris Buffered Saline (TBS) — One injection, solution for injection, intramuscular use, 0.5mL TBS, pH 7.7.
  Arms: Group 2: Single dose Placebo

SUMMARY:
Phase 3 randomized, double blind study comparing recombinant MVA-BN-RSV vaccine vs placebo for efficacy and safety in adults >=60 years of age

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥60 years of age.
2. Informed Consent signed by the subject.
3. Subjects may have one or more chronic medical conditions e.g., mild to moderate underlying illnesses such as chronic cardiac diseases and chronic lung disease (asthma and chronic obstructive pulmonary disease [COPD]), congestive heart failure (CHF), hypertension, type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism, that is clinically stable as assessed by the investigator.
4. Absence of known, current, and life-limiting diagnoses that render survival to completion of the protocol unlikely.
5. Ability to comply with trial requirements, which necessitates access to transportation to on-site visits, including symptom visits for a nasopharyngeal swab.
6. Willingness and ability to utilize an application on a personal device (i.e., smartphone, tablet, etc.) or a provisioned device to record solicited events and record all per protocol required data during the surveillance period.
7. For women of childbearing potential (WOCBP), agreement to use an acceptable method of contraception during the trial and a negative urine pregnancy test within 24 hours prior to vaccination.

Exclusion Criteria:

1. History of or current clinical manifestation of any serious medical condition that in the opinion of the investigator would compromise the safety of the subject, confound data interpretation, or would limit the subject's ability to complete the trial.
2. History of or active autoimmune disease, including diabetes mellitus type I. Vitiligo or hypothyroidism requiring thyroid replacement therapy are not exclusions. Rheumatoid arthritis not requiring immunomodulatory and/or immunosuppressant treatment is not an exclusion.
3. Known or suspected impairment of immunologic functions, including chronic inflammatory bowel disorders.
4. Clinically significant mental disorder that would prevent patients from giving informed consent and complying with study procedures (e.g., completion of the electronic diary).
5. Active or recent (within 6 months before enrollment) history of chronic alcohol abuse.
6. History of a serious reaction to any prior vaccination or Guillain-Barré syndrome (GBS) within 6 weeks of any prior influenza immunization.
7. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g., tris(hydroxymethyl)-amino methane, chicken embryo fibroblast proteins, gentamycin, ciprofloxacin; this includes:

   * Known allergy to eggs or aminoglycosides
   * History of anaphylaxis or severe allergic reaction to any vaccine
8. Any administration or planned administration of:

   * A licensed live or vector-based vaccine within 30 days prior to or after trial vaccine administration.
   * A licensed inactivated or ribonucleic acid (RNA)-based vaccine within 14 days prior to or after trial vaccine administration.
9. Previous vaccination with an RSV vaccine, or any planned vaccination with an RSV vaccine other than the trial vaccine.
10. Planned chronic, systemic administration (defined as more than 14 days) of >10 mg prednisone (or equivalent)/day or any other systemic use of immunemodifying drugs during a period starting from 3 months prior to first administration of the trial vaccine and ending at the End of Study Visit (EOS). The use of topical, inhaled, ophthalmic and nasal glucocorticoids is permitted.
11. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from 3 months prior to first administration of the trial vaccine and during the trial.
12. Known uncontrolled coagulation disorder. Anticoagulant treatment under adequate control for cardiovascular prophylaxis or prophylaxis of thromboembolic disease or stroke in the setting of atrial fibrillation are permitted.
13. Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days prior to the administration of the trial vaccine, or planned administration of such a drug or vaccine between enrollment in the trial and until the end of the clinical trial including follow-up. [For US Only]
14. Involvement with this trial as research personnel.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20419 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Hoet, MD, Study Director — Bavarian Nordic
Locations (120):
- United States (105):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Achieve Clinical Research, LLC d/b/a Accel Research Sites, Birmingham, Alabama
  - Medical Affiliation Research Center, Huntsville, Alabama
  - Lenzmeier Family Medicine / CCT Research, Glendale, Arizona
  - Aventiv Research Inc., Mesa, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - Pain Center of Arizona, Phoenix, Arizona
  - Cognitive Clinical Trials, LLC, Phoenix, Arizona
  - Fiel Family and Sports Medicine/CCT Research, Tempe, Arizona
  - HOPE Research Institute, Tempe, Arizona
  - Tucson Neuroscience Research, LLC, Tucson, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Hope Clinical Research, LLC, Canoga Park, California
  - Marvel Clinical Research 002, LLC, Huntington Beach, California
  - Join Clinical Trials, Huntington Park, California
  - Paradigm Clinical Research Center, La Mesa, California
  - Atella Clinical Research LLC, La Palma, California
  - Chemidox Clinical Trials Inc., Lancaster, California
  - ARK Clinical Research, Long Beach, California
  - Matrix Clinical Research, Los Angeles, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Research Foundation, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Innovative Research Of West Florida, Inc., Clearwater, Florida
  - Doral Medical Research, Hialeah, Florida
  - K2 Medical Research, LLC, Maitland, Florida
  - Optimus U Corporation, Miami, Florida
  - De La Cruz Research Center, LLC, Miami, Florida
  - Global Health Research Center, Inc, Miami Lakes, Florida
  - Pines Care Research Center, LLC, Pembroke Pines, Florida
  - IDEAL Clinical Research, Pembroke Pines, Florida
  - Centricity Research Columbus Multispecialty, Columbus, Georgia
  - Accel Research Site - Neurostudies, Decatur, Georgia
  - Lifeline Primary Care/CCT Research, Lilburn, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Great Lakes Clinical Trials at Ravenswood Rheumatology, Chicago, Illinois
  - Accelacare- DuPage Medical Group, Oak Lawn, Illinois
  - AES Evansville, Evansville, Indiana
  - Accellacare and McFarland Clinic, Ames, Iowa
  - Meridian Clinical Research, Sioux City, Iowa
  - Med Pharmics, LLC, Metairie, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - Meridian Clinical Research, Rockville, Maryland
  - ActivMed Practices and Research, LLC, Methuen, Massachusetts
  - Henry Ford Health Hospital, Detroit, Michigan
  - Edward A. Doisy Research Center-Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Meridian Clinical Research, LLC, Grand Island, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Quality Clinical Research Inc, Omaha, Nebraska
  - Meridian Clinical Research Associates, LLC, Omaha, Nebraska
  - Midwest Regional Health Services, LLC/CCT Research, Omaha, Nebraska
  - Synexus Clinical Research US, Inc., Henderson, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada/ CCT Research, Las Vegas, Nevada
  - Amici Clinical Research, Raritan, New Jersey
  - MedPharmics, LLC, Albuquerque, New Mexico
  - Certified Research Associates, Cortland, New York
  - Meridian Clinical Research LLC, Endwell, New York
  - CHEAR Center LLC, New York, New York
  - Rochester Clinical Research Inc., Rochester, New York
  - Accellacare - Raleigh Medical Group, Cary, North Carolina
  - Accellacare Research of Charlotte, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Accellacare - Raleigh Medical Group, Raleigh, North Carolina
  - Accellacare, Inc. - Rocky Mount, Rocky Mount, North Carolina
  - Accellacare - Piedmont, Statesville, North Carolina
  - Accellacare of Wilmington, Wilmington, North Carolina
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - Tekton Research, Moore, Oklahoma
  - Lynn Health Science Institute East, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Tekton Research Inc., Yukon, Oklahoma
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - DM Clinical Research, Philadelphia, Pennsylvania
  - Velocity Clinical Research- Providence, East Greenwich, Rhode Island
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Velocity Clinical Research Anderson, Anderson, South Carolina
  - Main Street Physician's Care-Waterway, Little River, South Carolina
  - Accellacare of Knoxville, Knoxville, Tennessee
  - Tekton Research, Inc., Austin, Texas
  - Invesclinic US LLC, Edinburg, Texas
  - DM Clinical Research, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Research Your Health, Plano, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Mt Olympus Medical Research LLC, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - Olympus Family Medicine/CCT Research, Holladay, Utah
  - Tanner Clinic, Layton, Utah
  - South Ogden Family Medicine/ CCT Research, Ogden, Utah
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Clinical Alliance for Research and Education Infectious Disease, Annandale, Virginia
  - Meridian Clinical Research, LLC, Portsmouth, Virginia
  - Centricity Research Suffolk Primary Care, Suffolk, Virginia
  - Sound Medical Research, Port Orchard, Washington
  - MultiCare Health System-DMOB (Deaconess Medical Office Building), Spokane, Washington
- Germany (15):
  - Klinische Forschung Berlin GbR, Berlin
  - Studienzentrum Diabetespraxis Dr. Braun, Berlin
  - MECS Cottbus GmbH, Cottbus
  - Klinsche Forschung Dresden GmbH, Dresden
  - IKF Institut fuer klinische Forschung Frankfurt, Frankfurt
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Siteworks GmbH, Hanover
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Siteworks Zentrum für Klinische Studien Heidelberg, Heidelberg
  - SIBAmed Studienzentrum GmbH & Co. KG, Leipzig
  - Dermatologische Gemeinschaftspraxis Dres. Quist, Mainz
  - RED Institut GmbH, Oldenburg
  - Siteworks Prufzentrum Rendsburg - HNO Research GmbH, Rendsburg
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Intermed GmbH, Institut fuer medizinische Forschung und Arzneimittelsicherheit, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jordan E, Jenkins V, Silbernagl G, Chavez MPV, Schmidt D, Schnorfeil F, Schultz S, Chen L, Salgado F, Jacquet JM, Welte T, De Moerlooze L. A multivalent RSV vaccine based on the modified vaccinia Ankara vector shows moderate protection against disease caused by RSV in older adults in a phase 3 clinical study. Vaccine. 2024 Dec 2;42(26):126427. doi: 10.1016/j.vaccine.2024.126427. Epub 2024 Oct 25. PMID 39461302

RESULTS

PARTICIPANT FLOW:
Groups:
- MVA-BN-RSV: Single administration of MVA-BN-RSV vaccine with a titer of at least 3 x 10E8 infectious units (Inf.U)/0.5mL (intramuscular injection).
  Group assignment based on the Full Analysis Set, i.e. participants randomized to MVA-BN-RSV and treated (including 8751 participants with a single randomization to MVA-BN-RSV [thereof 4 participants actually received Placebo] and 409 participants [multiple enrollers] with their first randomization to MVA-BN-RSV [thereof 230 participants receiving Placebo as second/later dose])
- Placebo: Single administration of Tris Buffered Saline (TBS) (intramuscular injection; 0.5mL).
  Group assignment based on the Full Analysis Set, i.e. participants randomized to Placebo and treated (including 8771 participants with a single randomization to Placebo [thereof 1 participant actually received MVA-BN-RSV] and 417 participants [multiple enrollers] with their first randomization to Placebo [thereof 232 participants receiving MVA-BN-RSV as second/later dose])
Period: Overall Study
Arm/Group | MVA-BN-RSV | Placebo
Started (Participants vaccinated) | 9160 | 9188
Completed (1 year follow-up) | 1530 | 1535
Not Completed | 7630 | 7653
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 334 | 339
Not completed — Withdrawal by Subject | 203 | 222
Not completed — Physician Decision | 20 | 8
Not completed — Protocol Violation | 6 | 2
Not completed — Death | 38 | 32
Not completed — Study terminated by Sponsor | 6358 | 6358
Not completed — Other Reason | 669 | 690

BASELINE CHARACTERISTICS:
Population: Full Analysis Set i.e., all participants who were randomized to any treatment arm and received study vaccine (MVA-BN-RSV or placebo). Participants were analyzed based on the treatment to which they were randomized. Participants who received multiple doses of study vaccine ("multiple enrollers") were included once in this analysis set with group allocation based on their first randomization.
Groups:
- MVA-BN-RSV: Single administration of MVA-BN-RSV vaccine with a titer of at least 3 x 10E8 infectious units (Inf.U)/0.5mL (intramuscular injection)
- Placebo: Single administration of Tris Buffered Saline (TBS) (intramuscular injection; 0.5mL)
- Total: Total of all reporting groups
Arm/Group | MVA-BN-RSV | Placebo | Total
Number analyzed (Participants) | 9160 | 9188 | 18348
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (5.78) | 70.5 (5.83) | 70.4 (5.81)
Age, Customized [Count of Participants; unit: Participants]
  60 to 64 years | 931 | 933 | 1864
  65 to 74 years | 6166 | 6164 | 12330
  75 to 84 years | 1889 | 1903 | 3792
  >= 85 years | 174 | 188 | 362
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4606 | 4680 | 9286
  Male | 4554 | 4508 | 9062
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7786 | 7794 | 15580
  Black or African American | 1185 | 1202 | 2387
  Asian | 79 | 63 | 142
  Native Hawaiian or Other Pacific Islander | 9 | 15 | 24
  American Indian or Alaska Native | 34 | 26 | 60
  Other | 67 | 87 | 154
  Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8445 | 8468 | 16913
  Germany | 715 | 720 | 1435

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of PCR Confirmed RSV-associated LRTD With at Least 3 Symptoms
Description: RSV-associated lower respiratory tract disease (LRTD) is defined by the presence of clinical evidence of at least 1 sign or symptom of acute respiratory disease (ARD) and at least 3 LRTD signs or symptoms with onset ≥14 days following vaccination until the end of one RSV season (up to 12 months after vaccination), confirmed and documented by a medical professional, together with RSV disease confirmed by polymerase chain reaction (PCR)
Time Frame: From 14 days post-vaccination up to the end of one RSV season, up to a maximum of 11 months
Population: Full Analysis Set i.e., all participants who were randomized to any treatment arm and received study vaccine (MVA-BN-RSV or placebo). Participants were analyzed based on the treatment to which they were randomized. Participants who received multiple doses of study vaccine ("multiple enrollers") were included once in this analysis set with group allocation based on their first randomization and with data censored from the time of second randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9160 | 9188
Participants | 12 | 21
Statistical Analysis 1: Comparison: MVA-BN-RSV vs Placebo; Test type: Other — Vaccine Efficacy (VE) is defined as 1 minus the hazard ratio resulting from a Cox proportional hazards regression model stratified by age group. It is demonstrated if the lower limit (LL) of the 2-sided 95% confidence interval (CI) for VE is above 20%; Vaccine Efficacy = 42.9, 95% CI 2-sided [-16.1 to 71.9]

2. Primary Outcome: Occurrence of PCR Confirmed RSV-associated LRTD With at Least 2 Symptoms
Description: RSV-associated lower respiratory tract disease (LRTD) is defined by the presence of clinical evidence of at least 1 sign or symptom of acute respiratory disease (ARD) and at least 2 LRTD signs or symptoms with onset ≥14 days following vaccination until the end of one RSV season (up to 12 months after vaccination), confirmed and documented by a medical professional, together with RSV disease confirmed by polymerase chain reaction (PCR)
Time Frame: From 14 days post-vaccination up to the end of one RSV season, up to a maximum of 11 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9160 | 9188
Participants | 25 | 61
Statistical Analysis 1: Comparison: MVA-BN-RSV vs Placebo; Test type: Other — Vaccine Efficacy (VE) is defined as 1 minus the hazard ratio resulting from a Cox proportional hazards regression model stratified by age group. It is demonstrated if the first primary outcome is met and the lower limit (LL) of the 2-sided 95% confidence interval (CI) for VE is above 20%; Vaccine Efficacy = 59.0, 95% CI 2-sided [34.7 to 74.3] — Not formally tested, since the first primary outcome was not met

3. Secondary Outcome: Occurrence of PCR Confirmed RSV-associated ARD
Description: RSV-associated acute respiratory disease (ARD) is defined by the presence of either one ARD symptom lasting for at least 24 hours or two simultaneously occurring ARD symptoms (irrespective of duration), with onset ≥14 days following vaccination until the end of one RSV season (up to 12 months after vaccination), confirmed and documented by a medical professional, together with RSV disease confirmed by polymerase chain reaction (PCR)
Time Frame: From 14 days post-vaccination up to the end of one RSV season, up to a maximum of 11 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9160 | 9188
Participants | 42 | 82
Statistical Analysis 1: Comparison: MVA-BN-RSV vs Placebo; Test type: Other — Vaccine Efficacy (VE) is defined as 1 minus the hazard ratio resulting from a Cox proportional hazards regression model stratified by age group. It is demonstrated if both primary outcomes are met and the lower limit (LL) of the 2-sided 95% confidence interval (CI) for VE is above 20%; Vaccine Efficacy = 48.8, 95% CI 2-sided [25.8 to 64.7] — Not formally tested, since the first primary outcome was not met

4. Secondary Outcome: Occurrence of Complications Related to PCR-confirmed RSV Disease
Description: RSV-specific complications include the presence of acute clinical consequences of RSV infection, such as pneumonia (incl. bacterial superinfection), sepsis, positive blood culture, and pneumothorax as well as longer term consequences of RSV-specific symptoms, such as persistent worsening of chronic conditions (e.g. COPD), new onset of persistent medical conditions (e.g. chronically impaired lung function, asthma) or a worsening of the functional status of the patient, e.g. new onset of nursing or assisted living need. RSV disease had to be confirmed by PCR testing.
Time Frame: From 14 days post-vaccination up to the end of one RSV season, up to a maximum of 11 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9160 | 9188
Participants | 0 | 1

5. Secondary Outcome: Occurrence of Hospitalization Due to Confirmed RSV Disease or Due to Any Complication Related to RSV-confirmed Respiratory Disease
Description: Hospitalization due to PCR confirmed RSV disease and/or any complication related to PCR-confirmed RSV disease. RSV-specific complications include the presence of acute clinical consequences of RSV infection, such as pneumonia (incl. bacterial superinfection), sepsis, positive blood culture, and pneumothorax as well as longer term consequences of RSV-specific symptoms, such as persistent worsening of chronic conditions (e.g. COPD), new onset of persistent medical conditions (e.g. chronically impaired lung function, asthma) or a worsening of the functional status of the patient, e.g. new onset of nursing or assisted living need. RSV disease had to be confirmed by PCR testing.
Time Frame: From 14 days post-vaccination up to the end of one RSV season, up to a maximum of 11 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9160 | 9188
Participants | 0 | 1

6. Secondary Outcome: Occurrence of Severe PCR Confirmed RSV-associated LRTD
Description: Severe RSV-associated LRTD is defined by the presence of clinical evidence of at least 1 sign or symptom of ARD and at least 1 of the following signs or symptoms with onset ≥14 days following vaccination until the end of one RSV season (up to 12 months after vaccination), confirmed and documented by a medical professional, together with RSV disease confirmed by polymerase chain reaction (PCR): 1) hypoxemia (oxygen saturation <92% at rest in conjunction with an at least 3% decrease from baseline); 2) respiratory rate >25 breaths/Min; 3) imaging evidence of new onset of bronchitis, bronchiolitis, or pneumonia
Time Frame: From 14 days post-vaccination up to the end of one RSV season, up to a maximum of 11 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9160 | 9188
Participants | 0 | 2

7. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Number and percentage of study participants reporting any serious adverse events at any time during the trial period.
Time Frame: From vaccination through study termination, up to 16 months
Population: Safety Set i.e., all participants who received study vaccine (MVA-BN-RSV or placebo). Subjects were analyzed based on the treatment they actually received. Subjects who received multiple doses of study vaccine ("multiple enrollers") were analyzed in the MVA-BN-RSV arm when having received the MVA-BN-RSV vaccine at least once; subjects were analyzed in the placebo arm when having received placebo only.
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9389 | 8959
Participants | 517 | 422

8. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Number and percentage of study participants reporting any grade 3 or higher unsolicited adverse events assessed as related to study vaccine
Time Frame: Within 29 days after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9389 | 8959
Participants | 11 | 2

9. Secondary Outcome: Number of Participants With Solicited Local Adverse Events
Description: Number and percentage of study participants reporting injection site reactions (solicited via electronic diaries) within 8 days after vaccination. The number of participants analyzed and the percentages are based on the subset of participants in the Safety Set that completed the electronic diary.
Time Frame: Within 8 days after vaccination
Population: Safety Set i.e., all participants who received study vaccine (MVA-BN-RSV or placebo). Subjects were analyzed based on the treatment they actually received. Subjects who received multiple doses of study vaccine ("multiple enrollers") were analyzed in the MVA-BN-RSV arm when having received the MVA-BN-RSV vaccine at least once; participants were analyzed in the placebo arm when having received placebo only.
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9389 | 8959
Participants
  Pain: number analyzed (Participants) | 9247 | 8829
  Pain | 5704 | 667
  Erythema: number analyzed (Participants) | 9247 | 8829
  Erythema | 522 | 157
  Swelling: number analyzed (Participants) | 9247 | 8829
  Swelling | 448 | 78
  Induration: number analyzed (Participants) | 9247 | 8829
  Induration | 417 | 74
  Pruritus: number analyzed (Participants) | 9247 | 8829
  Pruritus | 1718 | 470

10. Secondary Outcome: Number of Participants With Solicited Systemic Adverse Events
Description: Number and percentage of study participants reporting systemic reactions (solicited via electronic diaries) within 8 days after vaccination. The number of participants analyzed and the percentages are based on the subset of participants in the Safety Set that completed the electronic diary.
Time Frame: Within 8 days after vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9389 | 8959
Participants
  Pyrexia: number analyzed (Participants) | 9247 | 8829
  Pyrexia | 550 | 309
  Headache: number analyzed (Participants) | 9247 | 8829
  Headache | 3144 | 1737
  Myalgia: number analyzed (Participants) | 9247 | 8829
  Myalgia | 4558 | 1480
  Chills: number analyzed (Participants) | 9247 | 8829
  Chills | 1531 | 490
  Nausea: number analyzed (Participants) | 9247 | 8829
  Nausea | 990 | 551
  Fatigue: number analyzed (Participants) | 9247 | 8829
  Fatigue | 3526 | 1973

11. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Number and percentage of study participants reporting any unsolicited adverse events within 29 days after vaccination.
Time Frame: Within 29 days after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 9389 | 8959
Participants | 607 | 581

12. Secondary Outcome: RSV-specific T-cell Responses
Description: RSV-specific T-cell responses measured 1 week post vaccination in a subset of the study population
Time Frame: 1 week after vaccination
Reporting Status: Not Posted

13. Secondary Outcome: RSV-specific Serum IgG Antibody Titers
Description: Geometric Mean Titers (GMTs) based on RSV-specific Immunoglobulin G (IgG) Enzyme-linked Immunosorbent Assay (ELISA)
Time Frame: 2 weeks after vaccination
Population: Immunogenicity Analysis Set, a subset of the Full Analysis Set, including participants at designated clinical trial sites who signed the informed consent form for collection of serum samples. Number of participants analyzed represent the participants with antibody titer results available at the respective time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 309 | 317
Titer
  Baseline: number analyzed (Participants) | 306 | 314
  Baseline | 1510.6 [1386.4 to 1646.0] | 1590.1 [1468.3 to 1722.0]
  Week 2: number analyzed (Participants) | 295 | 290
  Week 2 | 4335.5 [3963.7 to 4742.2] | 1562.9 [1440.5 to 1695.6]

14. Secondary Outcome: RSV-specific Serum Neutralizing Antibody Titers (Subtype A)
Description: Geometric Mean Titers (GMTs) based on RSV-specific Plaque Reduction Neutralization Test (PRNT; against subtype A). Results below the lower limit of quantitation (LLOQ) are included with a value of 1/2 LLOQ
Time Frame: 2 weeks after vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 309 | 317
Titer
  Baseline: number analyzed (Participants) | 306 | 314
  Baseline | 275.1 [249.4 to 303.4] | 310.6 [280.5 to 343.9]
  Week 2: number analyzed (Participants) | 295 | 290
  Week 2 | 482.3 [436.9 to 532.5] | 307.7 [276.5 to 342.4]

15. Secondary Outcome: RSV-specific Serum Neutralizing Antibody Titers (Subtype B)
Description: Geometric Mean Titers (GMTs) based on RSV-specific Plaque Reduction Neutralization Test (PRNT; against subtype B). Results below the lower limit of quantitation (LLOQ) are included with a value of 1/2 LLOQ
Time Frame: 2 weeks after vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MVA-BN-RSV | Placebo
Number analyzed (Participants) | 309 | 317
Titer
  Baseline: number analyzed (Participants) | 306 | 314
  Baseline | 289.5 [251.5 to 333.1] | 336.5 [292.1 to 387.5]
  Week 2: number analyzed (Participants) | 295 | 290
  Week 2 | 475.3 [419.7 to 538.3] | 307.6 [265.4 to 356.5]

ADVERSE EVENTS:
Time Frame: From vaccination through study termination, up to 16 months
Description: SAEs were to be reported from vaccination to study end, non-serious AEs within 4 weeks of vaccination. Participants were analyzed based on their actual treatment. Multiple enrollers with at least 1 dose of MVA-BN-RSV were analyzed in the MVA-BN-RSV group from administration of MVA-BN-RSV onwards. Multiple enrollers receiving Placebo first and at least one dose of MVA-BN-RSV later were also analyzed in the Placebo group starting from administration of Placebo up to administration of MVA-BN-RSV.
Groups:
- MVA-BN-RSV: Single administration of MVA-BN-RSV vaccine with a titer of at least 3 x 10E8 infectious units (Inf.U)/0.5mL (intramuscular injection).
  Group assignment based on actual treatment, i.e. participants treated with MVA-BN-RSV (including 8747 Single Enroller participants randomized to MVA-BN-RSV and treated with MVA-BN-RSV + 1 Single Enroller participant randomized to Placebo and treated with MVA-BN-RSV + 179 Multiple Enroller participants randomized to MVA-BN-RSV (first randomization) and treated with MVA-BN-RSV only + 230 Multiple Enroller participants randomized to MVA-BN-RSV (first randomization) and treated with at least one dose of Placebo + 232 Multiple Enroller participants randomized to Placebo (first randomization) and treated with at least one dose of MVA-BN-RSV).
- Placebo: Single administration of Tris Buffered Saline (TBS) (intramuscular injection; 0.5mL).
  Group assignment based on actual treatment, i.e. participants treated with Placebo (including 8770 Single Enroller participants randomized to Placebo and treated with Placebo + 4 Single Enroller participants randomized to MVA-BN-RSV and treated with Placebo + 185 Multiple Enroller participants randomized to Placebo (first randomization) and treated with Placebo only (at least 2 doses and up to 4 doses) + 232 Multiple Enroller participants randomized to Placebo (first randomization) and treated with at least one dose of MVA-BN-RSV).
Arm/Group | MVA-BN-RSV | Placebo
All-Cause Mortality (participants affected / at risk) | 41/9389 | 34/9191
Serious Adverse Events (participants affected / at risk) | 517/9389 | 422/9191
Other Adverse Events (participants affected / at risk) | 82/9389 | 82/9191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MVA-BN-RSV (N=9389) | Placebo (N=9191)
Pneumonia (Infections and infestations) | 37 | 23
Sepsis (Infections and infestations) | 12 | 9
Cellulitis (Infections and infestations) | 10 | 6
COVID-19 (Infections and infestations) | 9 | 5
Urinary tract infection (Infections and infestations) | 9 | 7
Diverticulitis (Infections and infestations) | 6 | 1
Arthritis infective (Infections and infestations) | 5 | 1
Appendicitis (Infections and infestations) | 4 | 3
COVID-19 pneumonia (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 3 | 2
Pyelonephritis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 3 | 4
Abscess limb (Infections and infestations) | 2 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 2 | 2
Localised infection (Infections and infestations) | 2 | 1
Metapneumovirus pneumonia (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Complicated appendicitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Fournier's gangrene (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 1 | 1
Hepatitis A (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Norovirus infection (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 3
Cholecystitis infective (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
External ear cellulitis (Infections and infestations) | 0 | 1
Fungaemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 1
Infected bite (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 2
Scrotal cellulitis (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 21 | 14
Acute myocardial infarction (Cardiac disorders) | 15 | 6
Myocardial infarction (Cardiac disorders) | 11 | 13
Angina pectoris (Cardiac disorders) | 9 | 6
Cardiac failure congestive (Cardiac disorders) | 8 | 3
Cardiac arrest (Cardiac disorders) | 6 | 1
Cardiac failure (Cardiac disorders) | 6 | 2
Coronary artery disease (Cardiac disorders) | 6 | 6
Cardiac failure acute (Cardiac disorders) | 3 | 3
Arrhythmia (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmic storm (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 2
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 2
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 4
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 3
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 15 | 11
Transient ischaemic attack (Nervous system disorders) | 12 | 6
Syncope (Nervous system disorders) | 9 | 8
Encephalopathy (Nervous system disorders) | 3 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 2
Metabolic encephalopathy (Nervous system disorders) | 2 | 1
Myelopathy (Nervous system disorders) | 2 | 1
Presyncope (Nervous system disorders) | 2 | 0
Alcoholic seizure (Nervous system disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Basal ganglia stroke (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0
Paralysis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 3
Speech disorder (Nervous system disorders) | 1 | 0
Bell's palsy (Nervous system disorders) | 0 | 1
Cervical spinal cord paralysis (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Lacunar stroke (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 2
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Colitis (Gastrointestinal disorders) | 4 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 2
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 3
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 2
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery occlusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal retrolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 4
Femur fracture (Injury, poisoning and procedural complications) | 5 | 1
Hip fracture (Injury, poisoning and procedural complications) | 5 | 6
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 5
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 3
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 4
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 4
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Marginal zone lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-cardiac chest pain (General disorders) | 11 | 3
Death (General disorders) | 9 | 7
Chest discomfort (General disorders) | 2 | 0
Chest pain (General disorders) | 2 | 3
Gait disturbance (General disorders) | 2 | 0
Malaise (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 3
Cardiac death (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Calcinosis (General disorders) | 0 | 1
Dysplasia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 4
Hypertensive crisis (Vascular disorders) | 4 | 1
Aortic stenosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypertensive emergency (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 6
Thrombosis (Vascular disorders) | 2 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 2
Internal haemorrhage (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Depression (Psychiatric disorders) | 5 | 3
Mental status changes (Psychiatric disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Alcohol use disorder (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Substance use disorder (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 2
Nephrolithiasis (Renal and urinary disorders) | 4 | 6
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
End stage renal disease (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Mixed incontinence (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 5 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 2
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Endometrial thickening (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Lens dislocation (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Gastrointestinal stoma output increased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Device dislocation (Product Issues) | 1 | 0
Device failure (Product Issues) | 1 | 0
Device loosening (Product Issues) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Gallbladder operation (Surgical and medical procedures) | 0 | 1
Hip surgery (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MVA-BN-RSV (N=9389) | Placebo (N=9191)
COVID-19 (Infections and infestations) | 82 | 82

LIMITATIONS AND CAVEATS:
Study terminated after the first RSV season, since the first primary endpoint was not met

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT05238025/Prot_SAP_000.pdf